CLINICAL TRIAL: NCT05626270
Title: Human Factors Validation Testing for Over-the-Counter Use of the Erchonia® LunulaLaser™ OTC
Brief Title: Human Factors Testing for OTC Use of the Erchonia® LunulaLaser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R-FFS-OTC
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- LunulaLaser OTC (Other): The user will be presented with the device in its intended packaging as if receiving it at their place of employment. No additional information, instruction or training will be provided by the Study Observer, or any other individual associated with the study. The user will be left to work out how to operate the Erchonia LunulaLaser™ OTC as independently and naturally as possible without interference or influence from the Study Observer. While the user will have received the instructional information in the packaging as in intended use, he or she will not be instructed to use any of the information. It will be up to the user as to if or how he or she chooses to use that information to set up operation of the device as would occur under actual conditions of intended use.
  Interventions: Device: LunulaLaser OTC

INTERVENTIONS:
Device: LunulaLaser OTC — The LunulaLaser™ OTC is a nonthermal and non-invasive procedure designed to restore the growth of clear, healthy nails in clients with onychomycosis.

SUMMARY:
Human factors validation testing to assess the intended user's ability to correctly, safely, and effectively set-up, activate and operate the LunulaLaser™ OTC, to administer a treatment to a suitably qualified client, and to understand the information contained in the Erchonia LunulaLaser™ OTC Installation and Proper Use Reference Guide and box labeling.

DETAILED DESCRIPTION:
This study is an uncontrolled simulated-use human factors validation testing design to assess the intended user's ability to correctly, safely, and effectively set-up, activate and operate the LunulaLaser™ OTC, to administer a treatment to a suitably qualified client, and to understand the information contained in the Erchonia LunulaLaser™ OTC Installation and Proper Use Reference Guide and box labeling.

The study design is comprehensive in scope and conducted in a manner such that the results will be able to be generalized to the actual intended user and client population under intended conditions of actual use and be adequately sensitive to capture use errors arising from either the user interface design and/or the instructional and informative materials. Study data will be collected in a manner that will facilitate analysis of the root causes of use errors or problems during the testing.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Male or female.
* Currently employed at a nail salon, beauty salon and/or spa, fitness and wellness spa, or the like.
* In possession of qualification(s), current licensure(s), certification(s), and/or accreditation(s), as applicable, to perform their designated tasks at their place of employment, e.g., cosmetology degree, nail technician, esthetician, massage therapist etc.
* Voluntarily signed consent form.

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Erchonia Corporation, Melbourne, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LunulaLaser OTC
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LunulaLaser OTC
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.13 (10.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Human Factors
Description: The outcome measure identifies the number of subject users that were defined as a study "pass".
  A subject user is determined a study 'pass if the subject satisfactorily completes both the device setup and treatment procedure. If the subject user does not satisfactorily complete either one or both of device setup and/or treatment procedure the subject will be determined a study "fail".
Time Frame: Each study session was completed on a single day, for up to 120 minutes
Population: Number of subject users that were defined as a study "pass".
Measure: Number; unit: participants
Arm/Group | LunulaLaser OTC
Number analyzed (Participants) | 15
participants | 15

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | LunulaLaser OTC
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/70/NCT05626270/Prot_SAP_000.pdf